CLINICAL TRIAL: NCT07194421
Title: In-Use Tolerance & Efficacy Study Under Dermatological Control of Sunscreen in Adults With Atopic Dermatitis Skin
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4620A20230439
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD); SCORAD Index(15-25)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: Adult intended to use Sunscreen RV4620A RP2552 product
  Interventions: Other: Sunscreen RV4620A RP2552

INTERVENTIONS:
Other: Sunscreen RV4620A RP2552 — Dermo-cosmetic product, Broadspectrum Sunscreen RV4620A RP2552, very high protection product Instructions for product use given to the subjects: Apply before and during sun exposure, at least twice daily. During sun exposure, applications must be renewed as often as necessary, in particular after swimming, perspiring, towelling, in order to ensure a good protection. On days of bad weather, apply the product in the morning and at the beginning of the afternoon.

SUMMARY:
This study evaluates a broad-spectrum SPF50+ sunscreen on 42 adults with Atopic Dermatitis, measuring skin tolerance and barrier function.

The study includes several visits as follow :

* Visit 1: Inclusion (Day 1)
* Visit 2: Intermediate Visit (Day 8)
* Visit 3: End of Study (Day 22)

ELIGIBILITY:
Inclusion Criteria:

* Phototype: from I to VI.
* Sun Exposure: Adults anticipating at least 6 exposures of 2 hours each during the study.
* Swimming Sessions: Subjects planning at least 4 swimming sessions, with a minimum of 50% intending to swim twice in the sea and twice in a pool.
* Sensitive Skin: At least 50% of subjects report having sensitive skin.
* Health Insurance: Must be registered with health social security or health insurance.
* Informed Consent: Must have signed the written Informed Consent form (ICF) for study participation.
* Personal Information: Must certify the accuracy of personal information provided to the Investigator.
* Health Status: Considered a "healthy subject" by the Investigator (excluding SCORAD considerations).
* Women of Childbearing Potential: Must agree to use an effective contraceptive method throughout the study and for at least 1 month prior to the inclusion visit.

Criteria Related to Skin Condition:

* Atopic Dermatitis: Subject must present atopic dermatitis according to the U.K Working Party's Diagnostic Criteria for Atopic Dermatitis, with mild atopic dermatitis indicated by a SCORAD score of 15 to 25 (inclusive), determined by a dermatologist.
* Reactivity: Must be reactive to external irritative factors such as chlorine, sand, salt, and sweat.

Non-Inclusion Criteria:

Criteria Related to Population:

* Subjects who have participated in another clinical trial within the week before the inclusion visit, or for a longer period if deemed necessary by the Investigator.
* Subjects currently participating or planning to participate in another clinical trial during the study, either in the same or a different investigation center.

Criteria Related to Subject's Health:

* Subjects experiencing a flare of atopic dermatitis.
* Pregnant or breastfeeding women (for women of childbearing potential).
* Subjects with dermatological conditions that may interfere with study data or are considered hazardous by the Investigator (e.g., pityriasis versicolor, severe pigmentation disorders such as vitiligo, melasma, multiple lentigines, numerous or large congenital nevi).
* Subjects with a personal medical history that may interfere with study data or is incompatible with study requirements (except if required by the Sponsor, e.g., atopic dermatitis).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects will be recruited from the investigation centre's panel. They will be selected on the basis of inclusion and non inclusion criteria specific to the study and on their ability to comply with the constraints required by the protocol. They will be definitely included in the study after a specific interview and a clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Global tolerance assessment by the investigator | At the end of the study, after Last Patient Out, (after Day 22)
  Global tolerance of the product is assessed on the "tolerance population" which includes all the subjects who applied investigational product at least once.
  This assessment allows for attribution of one of the 5 levels : excellent, very good, good, moderate, bad.

SECONDARY OUTCOMES:
Evaluation Cosmetic Acceptability of the Sunscreen RV4620A - RP2552 | Visit 3 (Day 22)
  The subjects answer a 10-questions questionnaire about user satisfaction, texture, and overall experience with the product, providing insights into its appeal and usability.
Evaluation of Irritative Factors with Sunscreen RV4620A - RP2552 | Visit 1 (Day 1, before investigational product application) and Visit 3 (Day 22)
  The subjects answer a questionnaire regarding the irritative factors
Evaluation of Transepidermal Water Loss with Sunscreen RV4620A - RP2552 | Visit 1 (Day 1, before investigational product application) and Visit 3 (Day 22)
  Trans Epidermal Water Loss measurements are done with a Tewameter TM 300® by a trained technician in a room with controlled temperature and hygrometry. This measurement aims to assess the effect of the investigational product on transepidermal water loss to determine the product's impact on the skin's barrier function.
Assessment of Skin pH with Sunscreen RV4620A - RP2552 | Visit 1 (Day 1, before investigational product application) and Visit 3 (Day 22)
  Measurement of the skin pH is done using the COURAGE & KHAZAKA PH 900 PC Skin pH meter fitted with an Ingold electrode. The goal is to determine the product's respect of skin surface pH.
Assessment of the Lipidic Index Evolution with Sunscreen RV4620A - RP2552 | Visit 1 (Day 1, before investigational product application) and Visit 3 (Day 22)
  The quantity of sebum excreted to the skin surface is quantitatively evaluated with a Sebumeter SM 815 (Courage & Khazaka). The goal is to determine the product's respect of skin's barrier function and seboregulating effect

CONTACTS AND LOCATIONS:
Locations (1):
- Insight Research, Quatre Bornes, Mauritius, Mauritius